CLINICAL TRIAL: NCT01274819
Title: Dynamic Light Application to Prevent ICU Acquired Delirium
Acronym: DLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeroen Bosch Ziekenhuis (Other)
Responsible Party: Principal Investigator, K.S. Simons, Drs, Jeroen Bosch Ziekenhuis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DLA 2011
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Delirium; Confusion
Keywords: delirium; confusion
MeSH Terms: conditions — Delirium; Confusion | interventions — Dynamic Light Scattering

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dynamic light (Experimental): ICU patients exposed to dynamic light during ICU stay
  Interventions: Other: Dynamic Light
- Normal Light (No Intervention): control group is exposed to normal light during ICU stay

INTERVENTIONS:
Other: Dynamic Light — Dynamic Light Application (DLA) is a light application which exposes the subject in the room to a varying light intensity and light temperature during the day thus mimicking a natural daylight exposure.
  Other Names: Philips
  Arms: Dynamic light

SUMMARY:
Rationale: Delirium is a frequently encountered problem in ICU patients and leads to increased morbidity and mortality; Delirium in the ICU is associated with sleep deprivation which is among others caused by a disrupted circadian rhythm; Dynamic Light application aims at restoring a proper circadian rhythm by rhythmically alternating light intensity and has shown beneficial effects in sleep quality. Whether DLA improves sleep quality and reduces delirium incidence in ICU patients is not known

Goals/endpoints:

To evaluate the feasibility of dynamic light application in the ICU and to study the effects of dynamic light application on the incidence of delirium, duration of mechanical ventilation, the number of ICU and hospital days, and mortality in a mixed population of medical and surgical ICU patients. In a subgroup of patients with a high risk of developing delirium, markers of circadian rhythm, inflammation and brain damage and post ICU HRQoL will be assessed Study design: prospective randomized single centre trial Study population: adult ICU patients > 18 years old with an expected duration of stay of more than 24 hours Intervention: Patients will be randomized between Standard Care or Standard Care + DLA; When receiving standard care, normal lighting settings will be used in that patient room, which can be controlled by the medical personnel; In the rooms of patients randomized to the DLA group, DL is applied with a changing intensity during the day according to a fixed rhythm, which is regulated centrally. In addition when necessary, an intervention light can be used which can be operated in the patient room.

Study parameters/endpoints: incidence of delirium as measured by the CAM-ICU; duration of mechanical ventilation, ICU and total hospital mortality; ICU and hospital LOS; Serum levels of inflammatory markers and markers of brain damage, urinary levels of markers of circadian rhythm, data of HRQoL questionnaires and total light exposure in both groups

DETAILED DESCRIPTION:
STUDY DESIGN This is a prospective randomized, single centre trial. The proposed starting date is 01-july- 2011 and the duration of the study will be 15 months.

All ICU patients who are expected to have an ICU stay of more than 24 hours are potential eligible. On ICU admission, patients will be screened for eligibility. The patients' demographics, patients' health status, medication use, APACHE II score, SOFA score and admission diagnosis will be reported at baseline. Before recruitment and enrollment in the study, each patient and/or relative will be given full explanation of the study and will be informed that they are free to discontinue their participation in the study at any time.

When considered eligible, patients will be given a unique patient number in consecutive order and will be assigned to the treatment corresponding with this number. Patients will be randomized in a one-on-one fashion according to a computer generated randomization list between Standard Care and Standard Care + DLA. The randomization list will be kept at the data co-ordination centre.

All of the 20 patient rooms on the 2 ICU wards are equipped with a special lighting system. This lighting system can offer the standard basic lighting in the patient room, with a set intensity and light colour, or the DL setting which offers changing light conditions depending on the time of the day, following a rhythmic pattern. In addition, all rooms have a basic low-intensity orientation light, which is turned on during night-time in all rooms.

The switch between the two modes is regulated centrally on a control panel that is located in the nursing station and cannot be altered in the patient-room

1.1 Standard Care On admission, a full physical examination is performed and, when possible, a history taken. An ECG and chest x-ray, when not performed shortly before, will be done. In addition, blood will be drawn from the indwelling arterial catheter for haemoglobin, leucocyte and thrombocyte count, renal and liver function, electrolytes, arterial blood gas analysis, lactate and markers of inflammation (C-reactive protein, procalcitonin). Blood pressure, heart rate, fluid balance, oxygen saturation are measured continuously and automatically registered in our Patient Data Management System (PDMS). When considered necessary, ventilatory support is commenced or continued (post-operative patients) and additional hemodynamic measurements performed.

All patients will receive thromboprophylaxis, when no clear contraindications exist, and ulcer prophylaxis. When patients are intubated, they receive analgesic and often sedative medications for patient comfort. If patients are expected to receive mechanical ventilation for at least 48 hours, Selective Digestive Decontamination (SDD) prophylaxis is commenced, consisting of application of oral and gastrointestinal antibiotic suspension, administration of four days of i.v. antibiotics (cefotaxime) and surveillance cultures.

Twice daily at 0800hrs and 2000hrs, routine blood analysis consisting of arterial blood gas analysis, haemoglobin, leucocyte and thrombocyte electrolytes, renal function and markers of inflammation, is performed. When no clear contraindications exist, sedative infusions are interrupted every morning since this has proven to decrease length of mechanical ventilation (39). In addition, when considered feasible, an attempt is made to "wean" the patient off the mechanical ventilator. Protocol-guided early mobilisation is commenced as soon as possible, directed by dedicated physical therapists.

Level of sedation is monitored as part of daily care by nurses in all patients every two hours using the Richmond Agitation Sedation Scale (RASS). This scale divides levels of consciousness indicated by a number ranging from -5 (unarousable) to +4 (combative, see Appendix). Ideally, patients have a RASS of 0 (alert and calm) and sedation is titrated to achieve a RASS of -2 to 0. In addition, screening on the presence of delirium is done using the CAM-ICU every eight hours by well trained ICU nurses . As has been mentioned before, this method has been validated for use in ICU patients and is easy to use by non-psychiatric personnel. When the CAM-ICU is positive, delirium treatment is started according to our protocol (see Appendix).

Standard measures to prevent delirium among our patients include maintaining a proper day-and- night rhythm by promoting night-time sleep (reduction of light and noise disturbance and reduction of daytime sleep using daily activity programs and mobilisation. When patients have visual or auditive impairments, glasses and hearing aids are being used as much as possible. A clock is present in each ICU room and relatives are asked to bring photographs of them so that patients can have some sense of familiarity. Dosages of deliriogenic medications (anticholinergics, opiates, benzodiazepines) are reduced as much as possible however cannot be ruled out completely since benzodiazepines and opiates are often used for sedation and analgesia.

When a patient is randomized to receive the basic light setting, standard lighting is used, including the possibility of using a high intensity intervention light when performing interventions. The light switch in the room then offers three options: 1) main light on 2) main light off 3) intervention light on/off.

1.2 Standard Care + DLA In addition to standard care, inpatients who are randomized at receiving DLA, the light switch in that room is set to DLA, as soon as possible after the patient is installed and initial investigation and handlings (e.g. placing urinary catheter, a central venous line and/or arterial cannula) have been performed. When interventions are necessary, a high intensity intervention light can be turned on manually by physicians or nurses. The lighting operation panel in this room then offers only one option, i.e. intervention light on/off. A computer will log the use of the dynamic lighting system,

1.3 Assessment During the first 24 hours, the risk of developing delirium will be assessed using the validated PRE-DELIRIC score. When patients with have a risk of developing delirium ≥>40%, they will be defined as a high risk patient.

In all patients, the presence of delirium is assessed three times a day until death or discharge off the ICU or death on fixed times using the CAM-ICU. When patients are unconscious, either because of their illness or due to sedative medications, the CAM-ICU cannot be performed and delirium cannot be assessed. This will be recorded in the case-record form.

Since delirium is associated with the use of sedatives and opioids, 24-hour dosages of these medications will be recorded daily at 8 am. For a list of these medications, see appendix.

In addition, renal function, (plasma creatinine and urea), electrolytes (sodium, potassium, ionized calcium) haemoglobin, white blood cell count, procalcitonin) will be monitored daily until discharge of the ICU. Total hospital length of stay will be registered for all patients. Patients will be analyzed in an intention-to-treat principle.

To assess differences in light exposure between the two groups, light levels are measured in every patient room, close to the patient's head. Since daylight may also influence total light exposure and differences exist in daylight exposure of the different patient rooms (See appendix 3) differences between light exposures in different rooms will be analysed and associated to the primary endpoint.

In patients with a high risk of developing delirium 5 ml of blood will be drawn on day 1,3,5,7, 14,21 and 28 and will be stored at -80 degrees Celsius until analysis. In addition in these high risk patients, circadian rhythm derived biomarkers will be determined by means of urinary excretion collected in 3-hour urinary samples during 24 hours on day 7, 14,21, 28 and then once per 2 weeks. To determine pre-existent quality of life a validated Health Related Quality of Life questionnaire will be used.

1.4 randomisation, blinding and allocation of treatment Patients will be randomized in one-on one fashion according to a computer generated randomization list. The randomization list will be kept at the data co-ordination centre. Since blinding is impossible with dynamic light, patients and relatives, nurses and doctors are aware of the treatment arm.

1.5 Study procedures DLA will be applied in the DLA group. In all patients 5 ml of blood will be drawn within 24 hours after admission and stored. In high risk patients, an extra 5 ml of blood will be collected during the morning laboratory rounds on day 1, 3, 5, 7, 14, 21 and 28. Since all patients have an indwelling arterial line and blood is already collected this is not considered to be an additional burden for the patient. In total a maximum of ca. 35 millilitres of blood during a period of 28 days will be collected. In addition in high risk patients, 3 -hour urinary samples will be collected during 24 hours on day 7, 14, 21, 28 and than every week until discharge off the ICU. On our ICU, all patients have an indwelling urinary catheter. On admission, a validated QoL questionnaire will be handed over to the patient or his/her next of kin to determine the pre-existent QoL; after 3, 6 and 12 months a QoL questionnaire will be sent to the patient to determine the post ICU QoL.

Analysis will be performed on the whole group but also in a post-hoc analysis where the effect of DLA will be analysed per season of admission.

ELIGIBILITY:
Inclusion Criteria:

* ICU-patients >18 yrs old
* expected duration of stay > 24 hrs

Exclusion Criteria:

* life expectancy of <48 hrs on ICU admission
* necessity of prolonged deep sedation
* blindness
* inability to speak or understand dutch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2011-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
delirium outcome | duration of ICU stay(average duration 5 days)
  This is a composite endpoint of incidence of delirium during ICU stay, 28-day delirium free days (28-DFD) and 28-day ventilator free days (28-VFD)

SECONDARY OUTCOMES:
ICU length-of-stay and ICU mortality | duration of ICU stay, (average duration 5 days)
  ICU length-of-stay and ICU mortality
duration of mechanical ventilation | duration of ICU stay (average duration 5 days)
Hospital length-of-stay and hospital mortality | duration of hospital stay (average duration 14 days)
serum levels of inflammatory markers and markers of brain damage | duration of ICU stay (average duration 5 days)
  when patients are considered to be at high risk of developing ICU acquired delirium ( using a validated scoring system) blood samples will be drawn on days 1, 3, 5, 7, 14, 21, and 28 after inclusion in the study and stored at -80 degrees until analysis.
urinary levels of markers of circadian rhythm | duration of ICU stay (average duration 5 days)
  in a subgroup of long-stay ICU patients 3-hour urinary samples of cortisol and melatonin will taken during 24 hours to determine the circadian rhythm and the possible effect of DLA on this rhythm
data of Health-related Quality of Life (HrQoL) questionnaires | during ICU stay and 3, 6 and 12 months after ICU discharge
  3 and 6 months after ICU discharge, a validated HrQoL will be sent to patients homes to assess their QoL after the ICU stay and to detect differences between the DLA and reference group
Delirium-free days without coma in 28 days | 28 days
  To assess whether Dynamic Light not only influences incidence of delirium, but also duration of delirium, 28-day delirium free days without coma is used as a marker of duration of delirium. Patients who leave the ICU with a delirium (defined as a positive CAM-ICU score within 3 days of ICU discharge) will be followed on the wards using nurse charts and the delirium observation scale (DOS) to assess duration of delirium after ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: KS Simons, drs, Principal Investigator — Jeroen Bosch Hospital
Locations (1):
- Jeroen Bosch Hospital, 's-Hertogenbosch, Netherlands

REFERENCES:
- [Background] Peterson JF, Pun BT, Dittus RS, Thomason JW, Jackson JC, Shintani AK, Ely EW. Delirium and its motoric subtypes: a study of 614 critically ill patients. J Am Geriatr Soc. 2006 Mar;54(3):479-84. doi: 10.1111/j.1532-5415.2005.00621.x. PMID 16551316
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Thomason JW, Shintani A, Peterson JF, Pun BT, Jackson JC, Ely EW. Intensive care unit delirium is an independent predictor of longer hospital stay: a prospective analysis of 261 non-ventilated patients. Crit Care. 2005 Aug;9(4):R375-81. doi: 10.1186/cc3729. Epub 2005 Jun 1. PMID 16137350
- [Background] Ouimet S, Kavanagh BP, Gottfried SB, Skrobik Y. Incidence, risk factors and consequences of ICU delirium. Intensive Care Med. 2007 Jan;33(1):66-73. doi: 10.1007/s00134-006-0399-8. Epub 2006 Nov 11. PMID 17102966
- [Background] Pisani MA, Kong SY, Kasl SV, Murphy TE, Araujo KL, Van Ness PH. Days of delirium are associated with 1-year mortality in an older intensive care unit population. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1092-7. doi: 10.1164/rccm.200904-0537OC. Epub 2009 Sep 10. PMID 19745202
- [Background] Balas MC, Happ MB, Yang W, Chelluri L, Richmond T. Outcomes Associated With Delirium in Older Patients in Surgical ICUs. Chest. 2009 Jan;135(1):18-25. doi: 10.1378/chest.08-1456. Epub 2008 Nov 18. PMID 19017895
- [Background] Milbrandt EB, Deppen S, Harrison PL, Shintani AK, Speroff T, Stiles RA, Truman B, Bernard GR, Dittus RS, Ely EW. Costs associated with delirium in mechanically ventilated patients. Crit Care Med. 2004 Apr;32(4):955-62. doi: 10.1097/01.ccm.0000119429.16055.92. PMID 15071384
- [Background] Leslie DL, Marcantonio ER, Zhang Y, Leo-Summers L, Inouye SK. One-year health care costs associated with delirium in the elderly population. Arch Intern Med. 2008 Jan 14;168(1):27-32. doi: 10.1001/archinternmed.2007.4. PMID 18195192
- [Background] Devlin JW, Fong JJ, Howard EP, Skrobik Y, McCoy N, Yasuda C, Marshall J. Assessment of delirium in the intensive care unit: nursing practices and perceptions. Am J Crit Care. 2008 Nov;17(6):555-65; quiz 566. PMID 18978240
- [Background] Inouye SK, Bogardus ST Jr, Charpentier PA, Leo-Summers L, Acampora D, Holford TR, Cooney LM Jr. A multicomponent intervention to prevent delirium in hospitalized older patients. N Engl J Med. 1999 Mar 4;340(9):669-76. doi: 10.1056/NEJM199903043400901. PMID 10053175
- [Background] Vidan MT, Sanchez E, Alonso M, Montero B, Ortiz J, Serra JA. An intervention integrated into daily clinical practice reduces the incidence of delirium during hospitalization in elderly patients. J Am Geriatr Soc. 2009 Nov;57(11):2029-36. doi: 10.1111/j.1532-5415.2009.02485.x. Epub 2009 Sep 15. PMID 19754498
- [Background] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Background] Riker RR, Shehabi Y, Bokesch PM, Ceraso D, Wisemandle W, Koura F, Whitten P, Margolis BD, Byrne DW, Ely EW, Rocha MG; SEDCOM (Safety and Efficacy of Dexmedetomidine Compared With Midazolam) Study Group. Dexmedetomidine vs midazolam for sedation of critically ill patients: a randomized trial. JAMA. 2009 Feb 4;301(5):489-99. doi: 10.1001/jama.2009.56. Epub 2009 Feb 2. PMID 19188334
- [Background] Pandharipande PP, Pun BT, Herr DL, Maze M, Girard TD, Miller RR, Shintani AK, Thompson JL, Jackson JC, Deppen SA, Stiles RA, Dittus RS, Bernard GR, Ely EW. Effect of sedation with dexmedetomidine vs lorazepam on acute brain dysfunction in mechanically ventilated patients: the MENDS randomized controlled trial. JAMA. 2007 Dec 12;298(22):2644-53. doi: 10.1001/jama.298.22.2644. PMID 18073360
- [Background] Maldonado JR, Wysong A, van der Starre PJ, Block T, Miller C, Reitz BA. Dexmedetomidine and the reduction of postoperative delirium after cardiac surgery. Psychosomatics. 2009 May-Jun;50(3):206-17. doi: 10.1176/appi.psy.50.3.206. PMID 19567759
- [Background] Devlin JW, Roberts RJ, Fong JJ, Skrobik Y, Riker RR, Hill NS, Robbins T, Garpestad E. Efficacy and safety of quetiapine in critically ill patients with delirium: a prospective, multicenter, randomized, double-blind, placebo-controlled pilot study. Crit Care Med. 2010 Feb;38(2):419-27. doi: 10.1097/CCM.0b013e3181b9e302. PMID 19915454
- [Background] Han CS, Kim YK. A double-blind trial of risperidone and haloperidol for the treatment of delirium. Psychosomatics. 2004 Jul-Aug;45(4):297-301. doi: 10.1016/S0033-3182(04)70170-X. PMID 15232043
- [Background] Kalisvaart KJ, de Jonghe JF, Bogaards MJ, Vreeswijk R, Egberts TC, Burger BJ, Eikelenboom P, van Gool WA. Haloperidol prophylaxis for elderly hip-surgery patients at risk for delirium: a randomized placebo-controlled study. J Am Geriatr Soc. 2005 Oct;53(10):1658-66. doi: 10.1111/j.1532-5415.2005.53503.x. PMID 16181163
- [Background] Cooper AB, Thornley KS, Young GB, Slutsky AS, Stewart TE, Hanly PJ. Sleep in critically ill patients requiring mechanical ventilation. Chest. 2000 Mar;117(3):809-18. doi: 10.1378/chest.117.3.809. PMID 10713011
- [Background] Freedman NS, Gazendam J, Levan L, Pack AI, Schwab RJ. Abnormal sleep/wake cycles and the effect of environmental noise on sleep disruption in the intensive care unit. Am J Respir Crit Care Med. 2001 Feb;163(2):451-7. doi: 10.1164/ajrccm.163.2.9912128. PMID 11179121
- [Background] Weinhouse GL, Schwab RJ, Watson PL, Patil N, Vaccaro B, Pandharipande P, Ely EW. Bench-to-bedside review: delirium in ICU patients - importance of sleep deprivation. Crit Care. 2009;13(6):234. doi: 10.1186/cc8131. Epub 2009 Dec 7. PMID 20053301
- [Background] Shirani A, St Louis EK. Illuminating rationale and uses for light therapy. J Clin Sleep Med. 2009 Apr 15;5(2):155-63. PMID 19968050
- [Background] Van Someren EJ, Kessler A, Mirmiran M, Swaab DF. Indirect bright light improves circadian rest-activity rhythm disturbances in demented patients. Biol Psychiatry. 1997 May 1;41(9):955-63. doi: 10.1016/S0006-3223(97)89928-3. PMID 9110101
- [Background] Satlin A, Volicer L, Ross V, Herz L, Campbell S. Bright light treatment of behavioral and sleep disturbances in patients with Alzheimer's disease. Am J Psychiatry. 1992 Aug;149(8):1028-32. doi: 10.1176/ajp.149.8.1028. PMID 1353313
- [Background] Wilson LM. Intensive care delirium. The effect of outside deprivation in a windowless unit. Arch Intern Med. 1972 Aug;130(2):225-6. doi: 10.1001/archinte.130.2.225. No abstract available. PMID 5050558
- [Background] Keep P, James J, Inman M. Windows in the intensive therapy unit. Anaesthesia. 1980 Mar;35(3):257-62. doi: 10.1111/j.1365-2044.1980.tb05093.x. PMID 7396137
- [Background] Taguchi T, Yano M, Kido Y. Influence of bright light therapy on postoperative patients: a pilot study. Intensive Crit Care Nurs. 2007 Oct;23(5):289-97. doi: 10.1016/j.iccn.2007.04.004. Epub 2007 Aug 9. PMID 17692522
- [Background] Scheer FA, Buijs RM. Light affects morning salivary cortisol in humans. J Clin Endocrinol Metab. 1999 Sep;84(9):3395-8. doi: 10.1210/jcem.84.9.6102. PMID 10487717
- [Background] Anderson JL, Glod CA, Dai J, Cao Y, Lockley SW. Lux vs. wavelength in light treatment of Seasonal Affective Disorder. Acta Psychiatr Scand. 2009 Sep;120(3):203-12. doi: 10.1111/j.1600-0447.2009.01345.x. Epub 2009 Feb 3. PMID 19207131
- [Background] Riemersma-van der Lek RF, Swaab DF, Twisk J, Hol EM, Hoogendijk WJ, Van Someren EJ. Effect of bright light and melatonin on cognitive and noncognitive function in elderly residents of group care facilities: a randomized controlled trial. JAMA. 2008 Jun 11;299(22):2642-55. doi: 10.1001/jama.299.22.2642. PMID 18544724
- [Background] Cajochen C, Zeitzer JM, Czeisler CA, Dijk DJ. Dose-response relationship for light intensity and ocular and electroencephalographic correlates of human alertness. Behav Brain Res. 2000 Oct;115(1):75-83. doi: 10.1016/s0166-4328(00)00236-9. PMID 10996410
- [Background] Zeitzer JM, Dijk DJ, Kronauer R, Brown E, Czeisler C. Sensitivity of the human circadian pacemaker to nocturnal light: melatonin phase resetting and suppression. J Physiol. 2000 Aug 1;526 Pt 3(Pt 3):695-702. doi: 10.1111/j.1469-7793.2000.00695.x. PMID 10922269
- [Background] Viola AU, James LM, Schlangen LJ, Dijk DJ. Blue-enriched white light in the workplace improves self-reported alertness, performance and sleep quality. Scand J Work Environ Health. 2008 Aug;34(4):297-306. doi: 10.5271/sjweh.1268. Epub 2008 Sep 22. PMID 18815716
- [Background] Dijk DJ, Cajochen C. Melatonin and the circadian regulation of sleep initiation, consolidation, structure, and the sleep EEG. J Biol Rhythms. 1997 Dec;12(6):627-35. doi: 10.1177/074873049701200618. PMID 9406038
- [Background] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Background] Oostenbrink JB, Koopmanschap MA, Rutten FF. Standardisation of costs: the Dutch Manual for Costing in economic evaluations. Pharmacoeconomics. 2002;20(7):443-54. doi: 10.2165/00019053-200220070-00002. PMID 12093300
- [Background] Aurell J, Elmqvist D. Sleep in the surgical intensive care unit: continuous polygraphic recording of sleep in nine patients receiving postoperative care. Br Med J (Clin Res Ed). 1985 Apr 6;290(6474):1029-32. doi: 10.1136/bmj.290.6474.1029. PMID 3921096
- [Derived] Westerdijk K, Simons KS, Zegers M, Wever PC, Pickkers P, de Jager CPC. The value of the neutrophil-lymphocyte count ratio in the diagnosis of sepsis in patients admitted to the Intensive Care Unit: A retrospective cohort study. PLoS One. 2019 Feb 27;14(2):e0212861. doi: 10.1371/journal.pone.0212861. eCollection 2019. PMID 30811475
- [Derived] Simons KS, van den Boogaard M, Hendriksen E, Gerretsen J, van der Hoeven JG, Pickkers P, de Jager CPC. Temporal biomarker profiles and their association with ICU acquired delirium: a cohort study. Crit Care. 2018 May 25;22(1):137. doi: 10.1186/s13054-018-2054-5. PMID 29801516
- [Derived] Simons KS, Laheij RJ, van den Boogaard M, Moviat MA, Paling AJ, Polderman FN, Rozendaal FW, Salet GA, van der Hoeven JG, Pickkers P, de Jager CP. Dynamic light application therapy to reduce the incidence and duration of delirium in intensive-care patients: a randomised controlled trial. Lancet Respir Med. 2016 Mar;4(3):194-202. doi: 10.1016/S2213-2600(16)00025-4. Epub 2016 Feb 16. PMID 26895652